CLINICAL TRIAL: NCT02513745
Title: Refractive Outcomes Evaluation of the Verion Image Guided System + ORA System With VerifEye
Brief Title: Conventional Surgery vs. Verion/VerifEye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolina Eyecare Physicians, LLC (Other)
Collaborators: Science in Vision (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP 2014-003
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-01

CONDITIONS: Cataract; Astigmatism
Keywords: cataract; toric; phacoemulsification
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Conventional (Active Comparator): Surgeon's standard of care prior to getting VERION. Spherical power will be selected using the surgeon's preferred formula (Haigis, Holladay 2, Holladay, or other) and biometry method (IOL Master, Lenstar). Astigmatism correction will be planned using the surgeon's preferred keratometry method and calculator/nomogram to determine toric power and corneal incisions (i.e. Alcon toric calculator, Holladay toric calculator, Abbott Medical Optics (AMO) LRI calculator, etc). At time of surgery, axis of placement will be marked using blue ink marks. Corneal incisions will be made manually.
  Interventions: Device: Conventional
- Refractive Cataract Suite (Verion + ORA) (Active Comparator): Digital Surgical Planning and Positioning Tools + ORA System with VerifEye or VerifEye +. Spherical power of the IOL will be selected using the Verion Planner with the surgeon's preferred formula with an optimized A-constant (Haigis, Holladay 2, Holladay, or other). Both toric lenses and corneal incisions will be calculated with the Verion Planner using the Verion Reference Unit keratometry and white to white measurements, and Lenstar biometry. The VERION Digital Markers L and M will be used for axis of placement and confirmed using ORA System with VerifEye or VerifEye +.
  Interventions: Device: Refractive Cataract Suite (Verion + ORA)

INTERVENTIONS:
Device: Conventional — Routine cataract surgery by phacoemulsification before laser-assisted cataract surgery.
  Arms: Conventional
Device: Refractive Cataract Suite (Verion + ORA) — Laser-assisted cataract surgery with the digital surgical planning and positioning tools, and intraoperative aberrometry.
  Arms: Refractive Cataract Suite (Verion + ORA)

SUMMARY:
Nowadays cataract patient's expectations are closer to those of refractive surgery patients. Patients want to be spectacle independent. However, fifteen to twenty percent of cataract surgery patients have from 1.00 to 3.00 diopters (D) of corneal astigmatism which makes achieving spectacle independence unlikely in this patients unless the astigmatism is treated at the time of cataract surgery. Option to treat this astigmatism include corneal or limbal incisions (LRIs), the use of toric intraocular lenses (IOLs) or LASIK. Regardless of the treatment of choice to correct the astigmatism at time of cataract extraction, a treatment plan has to be calculated preoperatively. This planning include: keratometry measurements and the use of a calculator to estimate the treatment and orientation of IOL and/or placement of the LRIs.

New technology has been developed and is widely used. Among this technology, we have the VERION Image Guided System. This system encompasses a reference unit that takes a picture of the eye with the patient in the sitting position creating image of the patient's eye, capturing scleral vessels, limbus and iris features. It measures keratometry as well as the corneal diameter (limbus) and pupil size. The information captured is transferred automatically to its planner where IOL power calculation and astigmatism correction calculation are completed. Additionally, intraoperative wavefront aberrometry has been used in the last couple of years with increase success.

DETAILED DESCRIPTION:
Nowadays cataract patient's expectations are closer to those of refractive surgery patients. Patients want to be spectacle independent. However, fifteen to twenty percent of cataract surgery patients have from 1.00 to 3.00 diopters (D) of corneal astigmatism which makes achieving spectacle independence unlikely in this patients unless the astigmatism is treated at the time of cataract surgery.

Currently available treatments include corneal or limbal incisions, the use of toric intraocular lenses (IOLs) or LASIK. Limbal relaxing incisions (LRIs) are the most commonly used manual method Traditionally, LRIs have been made manually (with a surgical knife). With the introduction of femtosecond laser to assist during cataract surgery, a new alternative is available for creating corneal incisions. The stability of the LRIs and visual outcomes using toric IOLs have been shown.

Regardless of the treatment of choice to correct the astigmatism at time of cataract extraction, a treatment plan has to be calculated preoperatively. This planning include: keratometry measurements and the use of a calculator to estimate the treatment and orientation of IOL and placement of the LRIs.

Keratometry can be measured using a variety of devices including manual keratometers (i.e. Javal-Shiotz), automated keratometers, corneal topography, and optical biometry ( IOL master and Lenstar).

Once keratometry to be used has been selected, if the treatment of choice are LRIs, a calculator is used to determine the location and size of the LRI. Many nomograms have been developed; the choice of nomogram is the surgeon's prefer one, usually based on prior experience, and their preferred knife. LRIs calculators are available on line. Nomograms specify the location, length, size, and number of incisions based on the patient's age, the type of astigmatism, and the amount of astigmatism correction needed.

If a toric IOL has been chosen then planning the appropriate orientation of the toric IOL is accomplished by using online calculators. The calculator selects the optimal toric power and location based on the keratometry and the surgically induced astigmatism (SIA) values entered by the surgeon.

Intraoperatively, marking the eye and placing the incisions or aligning the toric IOL in the right axis are key steps for the success of astigmatism correction. Marking of the eye can be done using a variety of instruments using ink and it is routinely done with the patient in the upright position to avoid cyclorotation. Once patient is on the table in supine position, axis should be checked once again. Additional suggested methods to mark the eye include taking pictures preoperatively to identify anatomical landmarks similar to iris registration in refractive surgery. The use of iris registration during LASIK was introduced in 2008. Several publications have shown that patients undergoing wavefront-guided LASIK with iris recognition achieved better visual and refractive outcomes compared to conventional LASIK.

Recently, Alcon introduced VERION Image Guided System: Digital Surgical Planning and Positioning Tools. This system encompasses a reference unit that takes a picture of the eye with the patient in the sitting position creating a high-resolution digital image of the patient's eye, capturing scleral vessels, limbus and iris features. It measures keratometry as well as the corneal diameter (limbus) and pupil size. The information captured is then transferred automatically to the planner where additional information including target refraction, manifest refraction, axial length, anterior chamber depth, and lens thickness is entered for IOL power calculation and astigmatism correction planning. Astigmatism correction options include corneal incisions, toric IOL and a combination of both. Intraoperatively, The VERION Digital Marker displays patient information and images from the VERION Reference Unit. Additionally it positions all incision locations and assists with lens alignment in real time while accounting for the variable impact of cyclorotation and patient eye movement. In the OR, it displays a reticle that helps to align the IOL to the axis according the surgical plan. It also helps to position manual LRIs.

Intraoperative wavefront aberrometry has been used in the last couple of years to confirm spherical and toric power as well as lens position. The Optiwave Refractive Analysis (ORA) system can refract the eye in phakic, aphakic, and pseudophakic states at any time during cataract surgery and assists in IOL power selection and recommendations for toric IOL positioning before and after implantation as well as LRIs confirming the surgery plan calculated preoperatively. Furthermore, VerifEye, an ORA hardware upgrade, provides continuous assessment of the patient's eye allowing for more precise measurements; therefore, more accurate results and improved refractive outcomes and VerifEye +, the latest upgrade that provides streaming information on the refractive status and correct IOL positioning through the right ocular of the surgical microscope. This enables the surgeon to visualize all the information without having to look up at the monitor screen during the surgical procedure.

This new technology is an alternative to plan and treat astigmatism at the time of cataract surgery. It could make this treatment easier for less experience surgeons by facilitating the calculations and making the identification of the correct axis easier by reducing the need for manual marks.

The main objective of this study is to evaluate spherical and astigmatism outcomes post routine cataract surgery when the complete VERION Image Guided System packet + ORA System with VerifEye or VerifEye + are used in the treatment of pre-existing astigmatism using toric intraocular lens (IOL) or corneal incisions compared to the surgeon's standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing bilateral cataract extraction or refractive lens exchange with intraocular lens implantation and astigmatism correction.
* Willing and able to provide written informed consent for participation in the study
* Willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

* Severe preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, retinal detachment, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmos or macrophthalmos, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc.
* Uncontrolled diabetes.
* Use of any systemic or topical drug known to interfere with visual performance.
* Contact lens use during the active treatment portion of the trial.
* Any concurrent infectious/non infectious conjunctivitis, keratitis or uveitis.
* Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules
* Previous refractive surgery.
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or study device implantation or may interfere with the interpretation of study results.
* Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.
* Intraocular conventional surgery within the past three months or intraocular laser surgery within one month in the operated eye.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D Solomon, MD, Principal Investigator — Carolina Eyecare Physicians, LLC
Locations (1):
- Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 84 eyes of 42 patients were enrolled and started the study.
Units Other Than Participants: Eyes
Groups:
- Refractive Cataract Suite (Verion + ORA): Digital Surgical Planning and Positioning Tools + ORA System with VerifEye or VerifEye +. Spherical power of the IOL will be selected using the Verion Planner with the surgeon's preferred formula with an optimized A-constant (Haigis, Holladay 2, Holladay, or other). Both toric lenses and corneal incisions will be calculated with the Verion Planner using the Verion Reference Unit keratometry and white to white measurements, and Lenstar biometry. The VERION Digital Markers L and M will be used for axis of placement and confirmed using ORA System with VerifEye or VerifEye +.
  Verion: Laser-assisted cataract surgery with the digital surgical planning and positioning tools, and intraoperative aberrometry.
Period: Overall Study
Arm/Group | Conventional | Refractive Cataract Suite (Verion + ORA)
Started (Contralateral eye study. 42 subjects/84 eyes. Each subject had 1 eye (randomized) in each group.) | 42; 42 Eyes | 42; 42 Eyes
Completed (Contralateral eye study. 39 subjects/78 eyes. Each subject had 1 eye (randomized) in each group.) | 39; 39 Eyes | 39; 39 Eyes
Not Completed | 3; 3 Eyes | 3; 3 Eyes
Not completed — Criteria at time of surgery not met. | 3 | 3

BASELINE CHARACTERISTICS:
Population: A total of 39 patients were included in the analysis. Eyes of each participant were assigned to each group (Conventional and Refractive Cataract Suite (Verion + ORA); therefore the total is the same number in each group.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional | Refractive Cataract Suite (Verion + ORA) | Total
Number analyzed (Participants) | 39 | 39 | 39
Number analyzed (Eyes) | 39 | 39 | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.11 (6.79) | 67.11 (6.79) | 67.11 (6.79)
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 26 | 26 | 52
  Male | 13 | 13 | 26
Race (NIH/OMB) [Count of Units; unit: Eyes]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 37 | 37 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Eyes]
  United States | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Residual Refractive Cylinder
Description: This is the manifest refractive cylinder measured 3 months after surgery. Note that because cataract surgery has been performed, there is no associated baseline value.
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Conventional | Refractive Cataract Suite (Verion + ORA)
Number analyzed (Participants) | 39 | 39
Diopters | 0.28 (0.25) | 0.33 (0.37)

2. Secondary Outcome: Residual Mean Spherical Equivalent Refraction
Description: This is the mean of the spherical equivalent refraction (sphere + 0.5*cylinder) from each eye. Note that because cataract surgery has been performed, there is no associated baseline value.
Time Frame: Three months
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Conventional | Refractive Cataract Suite (Verion + ORA)
Number analyzed (Participants) | 39 | 39
Diopters | 0.06 (0.22) | 0.02 (0.31)

3. Secondary Outcome: Residual Corneal Astigmatism
Description: This is the anterior corneal astigmatism measured through keratometry. Note that because cataract surgery has been performed, there is no associated baseline value.
Time Frame: Three months
Population: This is a contra-lateral eye study where the first eye undergoing surgery was randomized to conventional or the refractive cataract suite, the fellow eye received the alternate treatment; therefore, we analyzed 78 eyes of 39 participants.
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Conventional | Refractive Cataract Suite (Verion + ORA)
Number analyzed (Participants) | 39 | 39
Diopters | 1.12 (0.71) | 1.16 (0.65)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the moment the participant signed the consent until exited the study that is about 4 months.
Arm/Group | Conventional | Refractive Cataract Suite (Verion + ORA)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 2/39 | 2/39
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional (N=39) | Refractive Cataract Suite (Verion + ORA) (N=39)
Irritation (Eye disorders) | 0 | 1
Worsening of dry eyes (Eye disorders) | 1 | 1
Retained lens fragments (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT02513745/Prot_SAP_000.pdf